CLINICAL TRIAL: NCT00882778
Title: Prophylactic Treatment With Recombinant Factor VIIa (rFVIIa, NovoSeven®) in Haemophilia Patients With Inhibitors
Brief Title: PROPACT: Retrospective Prophylaxis Patient Case Collection
Acronym: PROPACT
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: F7HAEM-3695
Record Dates: First submitted 2009-04-14; First posted 2009-04-16 (Estimated); Results first posted 2011-07-25 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A With Inhibitors; Haemophilia B With Inhibitors
MeSH Terms: interventions — Factor VII

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- activated recombinant human factor VII: Male patients diagnosed with haemophilia A or B with inhibitors, who were prescribed activated recombinant human factor VII (rFVIIa) for at least 30 days. All direction for rFVIIa medication usage was at the sole discretion of the physician in accordance within their usual practice. Data was collected for approximately 6 months of pre-prophylaxis, while the prophylaxis period had no limits.
  Interventions: Drug: eptacog alfa (activated)

INTERVENTIONS:
Drug: eptacog alfa (activated) — Retrospective data collection of the use of activated recombinant human factor VII as prophylaxis in haemophilia patients with inhibitors
  Other Names: activated recombinant human factor VII

SUMMARY:
This study is conducted in Europe and North and South America. The primary aim of this observational study is to evaluate the frequency and pattern of bleeding episodes in haemophilia patients receiving preventative treatment with activated recombinant human factor VII. The secondary aim is to evaluate which patients are selected for this treatment, the dose and dose intervals used, and the safety of activated recombinant human factor VII when used as prevention. The study also aims to increase understanding of the unmet medical need and clinical relevance of preventative treatment in haemophilia patients.

ELIGIBILITY:
Inclusion Criteria:

* Haemophilia A or B with inhibitors
* Prescribed use of activated recombinant human factor VII for any type of prophylaxis with a duration of at least 30 days

Exclusion Criteria:

* Prophylaxis prescribed post-surgery
* One or more coagulation disorders in addition to haemophilia

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Haemophilia patients in specialist hospital clinic or private clinic settings
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2009-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (14):
- Novo Nordisk Investigational Site, Princeton, New Jersey, United States
- Novo Nordisk Investigational Site, Prov. de Buenos Aires, Argentina
- Novo Nordisk Investigational Site, Mississauga, Canada
- Novo Nordisk Investigational Site, Zagreb, Croatia
- Novo Nordisk Investigational Site, Prague, Czechia
- Novo Nordisk Investigational Site, Paris La Défense Cedex, France
- Novo Nordisk Investigational Site, Mainz, Germany
- Novo Nordisk Investigational Site, Dublin, Ireland
- Novo Nordisk Investigational Site, Rome, Italy
- Novo Nordisk Investigational Site, Bratislava, Slovakia
- Novo Nordisk Investigational Site, Madrid, Spain
- Novo Nordisk Investigational Site, Malmo, Sweden
- Novo Nordisk Investigational Site, Zurich, Switzerland
- Novo Nordisk Investigational Site, Crawley, United Kingdom

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participating sites: Argentina (1), Canada (1), Croatia (1), Czech Republic (1), Germany (1), France (1), Ireland (1), Italy (4), Slovakia (1), Spain (3), Sweden (2), Switzerland (2), United Kingdom (1), and the United States of America (11)
Period: Overall Study
Arm/Group | Activated Recombinant Human Factor VII
Started | 86
Completed | 86
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 86
Age, Continuous [Mean (Standard Deviation); unit: years] — All = participants from bleeding population and frequent bleeding population (FBP). The FBP is a subset of the bleeding population with at least one bleed per month in the pre-prophylactic period of approximately 6 months.
  years
    All, n=86 | 11.6 (13.03)
    Bleeding population, n=74 | 10.9 (12.45)
    Frequent bleeding population, n=36 | 12.1 (12.67)
Age, Customized [Number; unit: participants]
  Below 12 years | 61
  Between 12 and 17 years | 7
  18 years or above | 18
Gender [Count of Participants; unit: Participants]
  Female | 0
  Male | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 7
  White | 43
  More than one race | 0
  Unknown or Not Reported | 33
Region of Enrollment [Number; unit: participants]
  Argentina | 4
  Canada | 1
  Croatia | 2
  Czech Republic | 1
  France | 17
  Germany | 3
  Ireland | 5
  Italy | 7
  Slovakia | 1
  Spain | 10
  Sweden | 4
  Switzerland | 2
  United Kingdom | 1
  United States | 28
Peak historical inhibitor titre recorded [Mean (Standard Deviation); unit: Bethesda Units (BU)/mL] — All = participants from bleeding population and frequent bleeding population (FBP). The FBP is a subset of the bleeding population with at least one bleed per month in the pre-prophylactic period of approximately 6 months.
  Bethesda Units (BU)/mL
    All, n=81 | 517.7 (1164.41)
    Bleeding population, n=72 | 571 (1224.88)
    Frequent bleeding population, n=35 | 737.9 (1457)
    Missing, n=5 | NA (NA) — No data available
Reason for prophylaxis [Number; unit: participants] — Reason patients were given prophylactic activated recombinant human factor VII
  participants
    Prevention of recurrent bleeding | 79
    In preparation for surgery | 0
    Prep. for rehab./planned phys. activity | 2
    Other | 2
    Missing | 3
Relationship to timing of Immune Tolerance Induction (ITI) [Number; unit: participants] — Timing (pre-, during, or post- Immune Tolerance Induction (ITI)) of prophylaxis determined within a subset of patients who had "prevention of recurrent bleeding" as the reason for prophylaxis
  participants
    Pre-ITI | 19
    During ITI | 8
    Post-ITI | 25
    ITI dates unknown | 0
    Not candidate for ITI | 27
    Not reported | 7
Duration of prophylaxis [Median (Full Range); unit: days] — All = participants from bleeding population and frequent bleeding population (FBP). The FBP is a subset of the bleeding population with at least one bleed per month in the pre-prophylactic period of approximately 6 months.
  days
    All, n=86 | 288 [22 to 3651]
    Bleeding population, n=74 | 293 [35 to 1580]
    Frequent bleeding population, n=36 | 293 [46 to 1580]
Weekly dose [Median (Full Range); unit: mcg/kg] — All = participants from bleeding population and frequent bleeding population (FBP). The FBP is a subset of the bleeding population with at least one bleed per month in the pre-prophylactic period of approximately 6 months.
  mcg/kg
    All, n=82 | 710 [94.2 to 3100]
    Bleeding population, n=73 | 742.5 [94.2 to 3100]
    Frequent bleeding population, n=36 | 656.2 [94.2 to 2768]
    Missing, n=4 | NA [NA to NA] — No data available
Dose frequency [Median (Full Range); unit: doses per week] — Average number of doses per week during prophylaxis period. All = participants from bleeding population and frequent bleeding population (FBP). The FBP is a subset of the bleeding population with at least one bleed per month in the pre-prophylactic period of approximately 6 months.
  doses per week
    All, n=82 | 5.2 [1 to 24.3]
    Bleeding population, n=73 | 5.8 [1 to 24.3]
    Frequent bleeding population, n=36 | 5.2 [1 to 22.2]
    Missing, n=4 | NA [NA to NA] — No data available

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Total Bleed Episodes Per Month - Bleeding Population
Description: Percent change of bleeds per month in the pre-prophylaxis period and bleeds per month in the prophylaxis period
Time Frame: Data was collected for an average of 6 months prior to start of prophylaxis (pre-prophylaxis period) and the period of prophylactic treatment (during prophylaxis), which had no time frame limits. Participants were on prophylaxis for a median of 288 days.
Population: Bleeding population with at least one bleed in the pre-prophylaxis period of approximately 6 months
Measure: Number; unit: percent change (%) in bleeds per month
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 74
percent change (%) in bleeds per month | -45

2. Primary Outcome: Percent Change in Total Bleed Episodes Per Month - Frequent Bleeding Population
Description: Percent change of bleeds per month in the pre-prophylaxis period and bleeds per month in the prophylaxis period
Time Frame: as for outcome 1
Population: Frequent bleeding population is a subset of patients in the bleeding population with at least one bleed per month in the pre-prophylaxis period of approximately 6 months
Measure: Number; unit: percent change (%) in bleeds per month
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 36
percent change (%) in bleeds per month | -51

3. Primary Outcome: Percent Change in Total Bleed Episodes Per Month Per Age Categories - Bleeding Population
Description: Percent change of bleeds per month between the pre-prophylaxis period and the prophylaxis period. Paediatric patients below 12 years, adolescents 12-17 years, and adults at least 18 years
Time Frame: as for outcome 1
Population: Bleeding population with at least one bleed in the pre-prophylaxis period of approximately 6 months
Measure: Number; unit: percent change (%) in bleeds per month
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 74
percent change (%) in bleeds per month
  Paediatric, n=54 | -48
  Adolescent, n=7 | 0
  Adult, n=13 | -56

4. Primary Outcome: Percent Change in Total Bleed Episodes Per Month Per Age Categories - Frequent Bleeding Population
Description: as for outcome 3
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number; unit: percent change (%) in bleeds per month
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 36
percent change (%) in bleeds per month
  Paediatric, n=27 | -56
  Adolescent, n=3 | 5
  Adult, n=6 | -49

5. Primary Outcome: Percent Change in Total Bleed Episodes Per Month by Dosing and Age Categories - Bleeding Population, Infrequent Dosing
Description: Percent change of bleeds per month between the pre-prophylaxis period and prophylaxis period. Paediatric patients below 12 years, adolescents 12-17 years, and adults at least 18 years. Infrequent dosing was defined as less than two doses per week. All participants = paediatrics, adolescents and adults.
Time Frame: as for outcome 1
Population: Bleeding population with at least one bleed in the pre-prophylaxis period of approximately 6 months
Measure: Number; unit: percent change (%) in bleeds per month
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 1
percent change (%) in bleeds per month
  All, n=1 | -6
  Paediatric, n=1 | -6
  Adolescent, n=0 | 0
  Adult, n=0 | 0

6. Primary Outcome: Percent Change in Total Bleed Episodes Per Month by Dosing and Age Categories - Bleeding Population, Dosing Three Times Per Week
Description: Percent change of bleeds per month between the pre-prophylaxis period and prophylaxis period. Paediatric patients below 12 years, adolescents 12-17 years, and adults at least 18 years. Three times per week dosing was defined as dosing two to four times per week. All participants = paediatrics, adolescents and adults.
Time Frame: as for outcome 1
Population: Bleeding population with at least one bleed in the pre-prophylaxis period of approximately 6 months
Measure: Number; unit: percent change (%) in bleeds per month
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 32
percent change (%) in bleeds per month
  All, n=32 | -52
  Paediatric, n=18 | -50
  Adolescent, n=3 | 12
  Adult, n=11 | -72

7. Primary Outcome: Percent Change in Total Bleed Episodes Per Month by Dosing and Age Categories - Bleeding Population, Daily Dosing
Description: Percent change of bleeds per month between the pre-prophylaxis period and prophylaxis period. Paediatric patients below 12 years, adolescents 12-17 years, and adults at least 18 years. Daily dosing was defined as 5 to 7 doses per week. All participants = paediatrics, adolescents and adults.
Time Frame: as for outcome 1
Population: Bleeding population with at least one bleed in the pre-prophylaxis period of approximately 6 months
Measure: Number; unit: percent change (%) in bleeds per month
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 29
percent change (%) in bleeds per month
  All, n=29 | -48
  Paediatric, n=26 | -48
  Adolescent, n=2 | -43
  Adult, n=1 | -51

8. Primary Outcome: Percent Change in Total Bleed Episodes Per Month by Dosing and Age Categories - Bleeding Population, Frequent Dosing
Description: Percent change of bleeds per month between the pre-prophylaxis period and the prophylaxis period. Paediatric patients below 12 years, adolescents 12-17 years, and adults at least 18 years. Frequent dosing was defined as 7 or more doses per week. All participants = paediatrics, adolescents and adults.
Time Frame: as for outcome 1
Population: Bleeding population with at least one bleed in the pre-prophylaxis period of approximately 6 months
Measure: Number; unit: percent change (%) in bleeds per month
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 11
percent change (%) in bleeds per month
  All, n=11 | -18
  Paediatric, n=8 | -47
  Adolescent, n=2 | 40
  Adult, n=1 | 35

9. Primary Outcome: Percent Change in Total Bleed Episodes Per Month by Dosing and Age Categories - Frequent Bleeding Population, Infrequent Dosing
Description: as for outcome 5
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number; unit: percent change (%) in bleeds per month
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 1
percent change (%) in bleeds per month
  All, n=1 | -6
  Paediatric, n=1 | -6
  Adolescent, n=0 | 0
  Adult, n=0 | 0

10. Primary Outcome: Percent Change in Total Bleed Episodes Per Month by Dosing and Age Categories - Frequent Bleeding Population, Dosing Three Times Per Week
Description: as for outcome 6
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number; unit: percent change (%) in bleeds per month
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 17
percent change (%) in bleeds per month
  All, n=17 | -56
  Padiatric, n=11 | -57
  Adolescent, n=2 | -10
  Adult, n=4 | -76

11. Primary Outcome: Percent Change in Total Bleed Episodes Per Month by Dosing and Age Categories - Frequent Bleeding Population, Daily Dosing
Description: as for outcome 7
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number; unit: percent change (%) in bleeds per month
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 15
percent change (%) in bleeds per month
  All, n=15 | -59
  Paediatric, n=13 | -62
  Adolescent, n=1 | 47
  Adult, n=1 | -51

12. Primary Outcome: Percent Change in Total Bleed Episodes Per Month by Dosing and Age Categories - Frequent Bleeding Population, Frequent Dosing
Description: Percent change of bleeds per month between the pre-prophylaxis period and prophylaxis period. Paediatric patients below 12 years, adolescents 12-17 years, and adults at least 18 years. Frequent dosing was defined as 7 or more doses per week. All participants = paediatrics, adolescents and adults.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number; unit: percent change (%) in bleeds per month
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 3
percent change (%) in bleeds per month
  All, n=3 | 33
  Paediatric, n=2 | -13
  Adolescent, n=0 | 0
  Adult, n=1 | 35

13. Secondary Outcome: Individual Dose by Dose Regimen and Age Group - Bleeding Population, Paediatric
Description: Individual activated recombinant human factor VII dose for paediatric patients by dosing regimen (infrequent dosing = less than 2 doses per week, three times per week = dosing 2-4 times per week, daily = 5-7 doses per week, or frequent dosing = 7 or more doses per week).
Time Frame: Data was collected for the period of prophylactic treatment (prophylaxis period), which had no time frame limits. Participants were on prophylaxis for a median of 288 days.
Population: Bleeding population with at least one bleed in the pre-prophylaxis period of approximately 6 months
Measure: Median (Full Range); unit: mcg/kg
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 53
mcg/kg
  Infrequent dosing, n=1 | 133.3 [133.3 to 133.3]
  Dosing three times per week, n=18 | 185.4 [26.9 to 301.8]
  Daily dosing, n=26 | 141.9 [54.5 to 395.4]
  Frequent dosing, n=8 | 135 [103.3 to 155.5]

14. Secondary Outcome: Individual Dose by Dose Regimen and Age Group - Bleeding Population, Adolescent
Description: Individual activated recombinant human factor VII dose for adolescent patients by dosing regimen (infrequent dosing = less than 2 doses per week, three times per week = dosing 2-4 times per week, daily = 5-7 doses per week, or frequent dosing = 7 or more doses per week).
Time Frame: as for outcome 13
Population: Bleeding population with at least one bleed in the pre-prophylaxis period of approximately 6 months
Measure: Median (Full Range); unit: mcg/kg
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 7
mcg/kg
  Infrequent dosing, n=0 | 0 [0 to 0]
  Dosing three times per week, n=3 | 198 [77.9 to 301.8]
  Daily dosing, n=2 | 138.9 [54.5 to 395.4]
  Frequent dosing, n=2 | 138 [120 to 155.5]

15. Secondary Outcome: Individual Dose by Dose Regimen and Age Group - Bleeding Population, Adult
Description: Individual activated recombinant human factor VII dose for adult patients by dosing regimen (infrequent dosing = less than 2 doses per week, three times per week = dosing 2-4 times per week, daily = 5-7 doses per week, or frequent dosing = 7 or more doses per week).
Time Frame: as for outcome 13
Population: Bleeding population with at least one bleed in the pre-prophylaxis period of approximately 6 months
Measure: Median (Full Range); unit: mcg/kg
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 13
mcg/kg
  Infrequent dosing, n=0 | 0 [0 to 0]
  Dosing three times per week, n=11 | 159.7 [26.9 to 290.9]
  Daily dosing, n=1 | 117.6 [117.6 to 117.6]
  Frequent dosing, n=1 | 103.3 [103.3 to 103.3]

16. Secondary Outcome: Individual Dose by Dose Regimen and Age Group - Frequent Bleeding Population, Paediatric
Description: as for outcome 13
Time Frame: as for outcome 13
Population: as for outcome 2
Measure: Median (Full Range); unit: mcg/kg
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 27
mcg/kg
  Infrequent dosing, n=1 | 133.3 [133.3 to 133.3]
  Dosing three times per week, n=11 | 197.2 [77.9 to 270]
  Daily dosing, n=13 | 135.9 [57.3 to 395.4]
  Frequent dosing, n=2 | 131 [127 to 135]

17. Secondary Outcome: Individual Dose by Dose Regimen and Age Group - Frequent Bleeding Population, Adolescent
Description: as for outcome 14
Time Frame: as for outcome 13
Population: as for outcome 2
Measure: Median (Full Range); unit: mcg/kg
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 3
mcg/kg
  Infrequent dosing, n=0 | 0 [0 to 0]
  Dosing three times per week, n=2 | 138 [96 to 180]
  Daily dosing, n=1 | 280 [280 to 280]
  Frequent dosing, n=0 | 0 [0 to 0]

18. Secondary Outcome: Individual Dose by Dose Regimen and Age Group - Frequent Bleeding Population, Adult
Description: as for outcome 15
Time Frame: as for outcome 13
Population: as for outcome 2
Measure: Median (Full Range); unit: mcg/kg
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 6
mcg/kg
  Infrequent dosing, n=0 | 0 [0 to 0]
  Dosing three times per week, n=4 | 162 [26.9 to 240]
  Daily dosing, n=1 | 117.6 [117.6 to 117.6]
  Frequent dosing, n=1 | 103.3 [103.3 to 103.3]

19. Secondary Outcome: Total Bleed Episodes Per Month by Joint, Target Joint and Non-joint - Bleeding Population
Description: Percent change in bleed episodes per month between pre-prophylaxis period and prophylaxis period by location of joint, target joint (defined as 3 or more documented bleeds in the same joint over the course of 6 months) or non-joint. All joints = target joints and non-target joints.
Time Frame: as for outcome 1
Population: Bleeding population with at least one bleed in the pre-prophylaxis period of approx. 6 months. Patients from the French sites were not included because bleed location was not collected. Bleed episodes with no recorded locations were not included in the analysis
Measure: Number; unit: percent change (%) in bleeds per month
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 56
percent change (%) in bleeds per month
  All joints | -39
  Target joints | -50
  Non-joints | -33

20. Secondary Outcome: Total Bleed Episodes Per Month by Joint, Target Joint and Non-joint - Frequent Bleeding Population
Description: Percent change in bleed episodes per month between pre-prophylaxis period and prophylaxis period by location of joint, target joint (= 3 or more documented bleeds in the same joint over the course of 6 months) or non-joint. All joints = target joints and non-target joints.
Time Frame: as for outcome 1
Population: Frequent bleeding population is a subset of patients in the bleeding population with at least one bleed per month in the pre-prophylaxis period of approx. 6 months. Patients from the French sites were not included because bleed location was not collected in these patients. Bleed episodes with no recorded locations were not included in the analysis
Measure: Number; unit: percent change (%) in bleeds per month
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 27
percent change (%) in bleeds per month
  All joints | -46
  Target joints | -56
  Non-joints | -42

21. Secondary Outcome: Healthcare Resource Consumption of Visits, Consultations, and Hospital Admissions Per Month - All Patients
Description: Healthcare resource consumption evaluated the absolute change in number of outpatient clinical visits, physician consultations and hospital admissions during the pre-prophylaxis to the prophylaxis period.
Time Frame: as for outcome 1
Population: Whole population of all male patients diagnosed with haemophilia A or B with inhibitor, who were prescribed activated recombinant human factor VII (rFVIIa) for at least 30 days
Measure: Mean (Standard Deviation); unit: change in events per month
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 83
change in events per month
  Out patient clinical visits | -0.011 (1.07)
  Physician consultations | 0.043 (1.66)
  Hospital admissions | -0.097 (0.27)

22. Secondary Outcome: Healthcare Resource Consumption of Visits, Consultations and Hospital Admissions Per Month - Bleeding Population
Description: Healthcare resource consumption evaluated the absolute change in number of outpatient clinical visits, physician consultations and hospital admissions during the pre-prophylaxis period to the prophylaxis period.
Time Frame: as for outcome 1
Population: Bleeding population with at least one bleed in the pre-prophylaxis period of approximately 6 months
Measure: Mean (Standard Deviation); unit: change in events per month
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 74
change in events per month
  Out patient clinical visits | 0.0090 (1.117)
  Physician consultations | 0.053 (1.76)
  Hospital admissions | -0.11 (0.28)

23. Secondary Outcome: Healthcare Resource Consumption of Visits, Consultations and Hospital Admissions Per Month - Frequent Bleeding Population
Description: as for outcome 22
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: change in events per month
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 36
change in events per month
  Out patient clinical visits | 0.0576 (1.39)
  Physician consultations | 0.213 (2.49)
  Hospital admissions | -0.11 (0.33)

24. Secondary Outcome: Healthcare Resource Consumption of Total Hospital Length of Stay and School/Work Absences Per Month - All Patients
Description: Healthcare resource consumption evaluated the absolute change in number of total hospital length of stay and school/work absences during the pre-prophylaxis period to the prophylaxis period.
Time Frame: as for outcome 1
Population: Whole population of all male patients diagnosed with haemophilia A or B with inhibitors, who were prescribed activated recombinant human factor VII (RFVIIa) for at least 30 days.
Measure: Mean (Standard Deviation); unit: change in days per month
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 83
change in days per month
  Total hospital length of stay | -0.654 (3.43)
  School/work absences | -1.365 (1.99)

25. Secondary Outcome: Healthcare Resource Consumption of Total Hospital Length of Stay and School/Work Absences Per Month - Bleeding Population
Description: as for outcome 24
Time Frame: as for outcome 1
Population: Bleeding population with at least one bleed in the pre-prophylaxis of approximately 6 months.
Measure: Mean (Standard Deviation); unit: change in days per month
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 74
change in days per month
  Total hospital length of stay | -0.794 (3.55)
  School/work absences | -1.365 (1.99)

26. Secondary Outcome: Healthcare Resource Consumption of Total Hospital Length of Stay and School/Work Absences Per Month - Frequent Bleeding Population
Description: as for outcome 24
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: change in days per month
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 36
change in days per month
  Total hospital length of stay | -1.064 (2.38)
  School/work absences | -1.927 (2.29)

27. Secondary Outcome: Physician Reported Outcome Assessment in Prophylaxis in Number of Patients
Description: Physician's assessment of prophylaxis outcome as successful, partially successful, unsuccessful, or unable to determine
Time Frame: as for outcome 1
Population: as for outcome 21
Measure: Number; unit: patients
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 86
patients
  Successful | 35
  Partially successful | 20
  Unsuccessful | 7
  Unable to determine | 9
  Data missing or not reported | 15

28. Secondary Outcome: Number of Physician Reported Outcome Assessment in Prophylaxis in Percentage of Patients
Description: Physician's assessment of prophylaxis outcome as successful, partially successful, unsuccessful, or unable to determine
Time Frame: as for outcome 1
Population: as for outcome 21
Measure: Number; unit: percentage of patients
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 86
percentage of patients
  Successful | 40
  Partially successful | 23
  Unsuccessful | 8
  Unable to determine | 10
  Data missing or not reported | 17

ADVERSE EVENTS:
Time Frame: Onset date 15-Dec-2007, outcome date 22-Dec-2007
Description: Safety population is all patients in the study. This is a non-interventional study, and thus only adverse events (AEs) and serious adverse events (SAEs) reported by the investigator is possible or probably related to drug and/or medical events of special interest (MESI) are included in the table
Arm/Group | Activated Recombinant Human Factor VII
Serious Adverse Events (participants affected / at risk) | 1/86
Other Adverse Events (participants affected / at risk) | 0/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Activated Recombinant Human Factor VII (N=86)
Septicaemia of Candida albicans (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No